CLINICAL TRIAL: NCT03712098
Title: Glucagon-like Peptide-1 Receptor Agonists as Novel Pharmacotherapies for Nicotine Dependence
Brief Title: Daily Liraglutide for Nicotine Dependence
Acronym: DAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rebecca Ashare (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Rebecca Ashare, Assistant Professor, Department of Psychiatry, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 831835
Record Dates: First submitted 2018-10-11; First posted 2018-10-19 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Smoking Cessation; Weight, Body
MeSH Terms: conditions — Smoking Cessation; Body Weight | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, parallel arm pilot study with one between-subjects factor of medication group (liraglutide vs. placebo).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smoking Cessation Counseling & Liraglutide (Experimental): Participants receive 8 sessions of smoking cessation behavioral counseling and 32 weeks of the medication liraglutide. Liraglutide comes in a pre-filled pen and is self-injected one time per day into the abdomen, thigh, or upper arm area. The dosing regimen, which follows FDA guidelines and is documented to be safe and well-tolerated in prior clinical studies, will begin at 0.6 mg and increase weekly by 0.6 mg until the recommended dose of 3 mg is reached (Weeks 1 through 5) and will continue at the 3 mg dose through the end of the study (Week 32).
  Interventions: Drug: Liraglutide; Behavioral: Smoking Cessation Counseling
- Smoking Cessation Counseling & Placebo (Active Comparator): Participants receive 8 sessions of smoking cessation behavioral counseling and 32 weeks of placebo. The placebo comes in a pre-filled pen and is self-injected one time per day into the abdomen, thigh, or upper arm area. The dosing regimen, which is the same as the liraglutide regimen, will begin at 0.6 mg and increase weekly by 0.6 mg until 3 mg is reached (Weeks 1 through 5) and will continue at the 3 mg dose through the end of the study (Week 32).
  Interventions: Drug: Placebo; Behavioral: Smoking Cessation Counseling

INTERVENTIONS:
Drug: Liraglutide — Liraglutide 3.0 mg is an injectable medicine that may help some adults with excess weight (BMI ≥27) who also have weight-related medical problems or obesity (BMI ≥30) lose weight and keep the weight off. Liraglutide is approved by the U.S. Food and Drug Administration (FDA) for chronic weight management when combined with a reduced-calorie meal plan and physical activity.
  Other Names: Saxenda
  Arms: Smoking Cessation Counseling & Liraglutide
Drug: Placebo — The placebo is an inactive substance that is designed to look like liraglutide but contains no medication.
  Arms: Smoking Cessation Counseling & Placebo
Behavioral: Smoking Cessation Counseling — All participants receive manual-based counseling from a trained smoking cessation counselor. The counseling sessions are designed to enhance awareness of the harmful effects of smoking, assist the participant in developing skills to quit, and avoid relapse.

SUMMARY:
This clinical research trial examines the effects of the GLP-1 receptor agonist liraglutide on smoking behavior, food intake, and weight gain. In this double-blind, placebo-controlled, parallel arm pilot study, overweight and obese smokers (N=40; 20 female and 20 male) will be randomized to 32 weeks of liraglutide or placebo and undergo 8 sessions of smoking cessation behavioral counseling. Outcomes are smoking abstinence and weight change.

DETAILED DESCRIPTION:
Tobacco use and obesity are the two leading causes of preventable deaths. A growing literature indicates that common neurobiological substrates mediate drug addiction and obesity. Therefore, it is not surprising that during smoking abstinence, highly palatable food may serve as a substitute reinforcer ultimately leading to increased body weight gain. Importantly, post-cessation weight gain (PCWG) can deter a quit attempt, precipitate smoking relapse, and contribute to health issues related to excess body weight. The majority of weight gain occurs within 3-6 months of quitting smoking and many individuals maintain this increased weight 5 to 20 years post-cessation. Although there is substantial variability in the amount of weight gained, individuals who successfully quit smoking gain an average of 4.2 kg, with estimates ranging from 2.5 kg to 8.6 kg, at 6-month follow-up. Weight gain after smoking cessation contributes to increased risk of obesity, type II diabetes mellitus and hypertension (18), as well as reducing the improvement in lung function conferred by smoking cessation. Moreover, overweight or obese smokers comprise 70% of treatment-seeking smokers, gain the most weight, and are the least accepting of PCWG. Thus, post-cessation weight gain is a significant clinical problem. Unfortunately, current pharmacological interventions to reduce post-cessation weight gain are not very effective.

While weight gain is often cited as a primary reason for smoking relapse, there is a significant gap in our understanding of the biobehavioral mechanisms linking smoking cessation and overeating. Recent evidence indicates that glucagon-like peptide-1 (GLP-1) regulates the rewarding effects of nicotine. These effects are mediated, in part, by reduced dopamine signaling in the nucleus accumbens, a key brain region known to regulate the reinforcing effects of both drugs of abuse and palatable foods. Indeed, activation of GLP-1 receptors in the ventral tegmental area (VTA), a brain region that sends dopaminergic projections to the nucleus accumbens, reduces both drug intake and consumption of palatable food. Based on the ability of GLP-1 receptor agonists to reduce drug and food intake, it is plausible that targeting GLP-1 receptor signaling may be an effective strategy toward reducing withdrawal-induced weight gain in abstinent smokers.

Investigators have recently developed a novel animal model of nicotine withdrawal-induced hyperphagia and body weight gain in order to gain an improved understanding of the molecular and behavioral mechanisms underlying increased food intake and body weight gain during nicotine withdrawal. The pilot data provide strong empirical rationale for the proposed study by establishing an animal model of withdrawal-induced hyperphagia and body weight gain following voluntary nicotine self-administration. This withdrawal phenotype was evident only in rats given ad libitum access to a highly palatable diet during withdrawal as parallel studies using a normal chow diet did not produce hyperphagia or changes in body weight during nicotine withdrawal (data not shown). Collectively,these results are consistent with human laboratory studies indicating that nicotine withdrawal is associated with increased consumption of highly palatable foods and body weight. The translational implications of studying this behavioral phenotype are clear and significant and include: 1) informing clinical approaches to treating weight gain during smoking abstinence, 2) identifying potential biomarkers associated with nicotine addiction, and 3) addressing two significant public health concerns.

GLP-1 receptor ligands are currently FDA-approved for the treatment of type II diabetes mellitus and obesity. Re-purposing an existing FDA-approved treatment that has been "de-risked" (i.e., previously shown to be safe) in numerous clinical trials removes a key barrier for drug development and reduces the resources required to bring new drugs to market.

The promising preclinical data, combined with evidence that GLP-1 receptor agonists are effective treatments for obesity, suggest that GLP-1 receptor ligands could be re-purposed for attenuating nicotine withdrawal-induced bodyweight gain, thereby improving smoking cessation rates. Specifically, this study will examine the effects of the GLP-1 receptor agonist liraglutide on smoking behavior as well as food intake and body weight gain during abstinence.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects will be males and females:

1. 18 years of age or older who self-report smoking cigarettes (menthol and non-menthol) at least 10 times per day, on average, for the past 6 months.
2. Interested in quitting smoking (defined as "intend to quit within one month").
3. Body mass index (BMI) greater than or equal to 27 kg/m2 with one weight-related comorbidity (e.g. high blood pressure, high cholesterol, dyslipidemia) or greater than or equal to 30 kg/m2 per the manufacturer label for weight management.
4. Women of childbearing potential (based on medical history) must consent to use a medically accepted method of birth control (e.g., condoms and spermicide, oral contraceptive, Depo-Provera injection, contraceptive patch, intrauterine device (IUD), tubal ligation) or agree to abstain from sexual intercourse during the time they are in the study.
5. Able to communicate (speak, read, and write) fluently in English.
6. Capable of giving written informed consent before any study-related activities, which includes compliance with the requirements and restrictions listed in the combined consent/HIPAA form.
7. If current or past diagnosis of bipolar disorder, eligible if:

   1. No psychotic features
   2. MADRS: total score less than 8 (past 4 weeks); suicidal item score less than 1 (past 4 weeks)
   3. Young Mania Rating Scale (Y-MRS): total score less than 8 (past 4 weeks); irritability, speech content, disruptive or aggressive behavior items score less than 3 (past 4 weeks)
   4. No psychiatric hospitalization or Emergency Room visits for psychiatric issues in the past 6 months
   5. No aggressive or violent acts or behavior in the past 6 months

Exclusion Criteria:

Subjects who present with and/or self-report the following criteria will not be eligible to participate in the study.

Smoking Behavior:

1. Current enrollment in a smoking cessation program, or use of other smoking cessation medications (e.g. Chantix/varenicline, Zyban/bupropion, nicotine replacement therapy/gum/patch, etc.) in the last month or plans to do either in the next 2 months.
2. Daily use of chewing tobacco, snuff and/or snus, or electronic cigarettes.

Alcohol/Drug Use:

1. Self-report current alcohol consumption that exceeds 25 standard drinks/week over the past 6 months.
2. Current untreated and unstable diagnosis of severe substance use disorder (eligible if past use and/or if receiving treatment and stable for at least 30 days). Current untreated and unstable moderate substance use disorder requires Study Physician approval.
3. A positive urine drug screen for cocaine, methamphetamines, phencyclidine (PCP), barbiturates, and/or ecstasy (MDMA).

   1. Participants believed to have a false-positive result on the drug screen may continue with the study with investigator approval.

Medical:

1. Females who self-report current pregnancy, planning a pregnancy during the study, currently breastfeeding/lactating, or not using adequate contraceptive measures. All female participants will undergo a urine pregnancy test at Intake and at every in-person study visit.
2. Current diagnosis of unstable and untreated major depression, as determined by self-report & MINI International Neuropsychiatric Interview (MINI) (eligible if stable for at least 30 days).
3. Current or past diagnosis of psychotic disorder, as determined by self-report or MINI. Mood Disorder with Psychotic Features determined by MINI requires PI approval for eligibility.
4. Suicide risk on the Columbia Suicide Severity Rating Scale (C-SSRS) indicated by active suicidal ideation (within past 30 days), any suicidal attempt within the past 2 years, or 2 or more lifetime suicidal attempts.
5. Self-reported kidney and/or liver disease or transplant.
6. Heart/Cardiovascular disease (e.g., angina, coronary heart disease, stroke, etc.) in the past 6 months.
7. Type-1 or type-2 diabetes (previously diagnosed or indicated by HbA1c level of 6.5% or higher).
8. Uncontrolled hypertension (BP systolic greater than 159 and/or diastolic greater than 99)*.
9. Personal or family history of medullary thyroid carcinoma (MTC).
10. Personal or family history of Multiple Endocrine Neoplasia syndrome type 2 (MEN 2).
11. History of pancreatitis.
12. History of gallbladder disease.
13. A blood glucose level less than 70 mg/dl at the Intake Visit.
14. Prior history, or plans, of surgical intervention for weight loss.
15. Hypersensitivity to liraglutide or any product components.
16. Current diagnosis of hyperthyroidism or hypothyroidism (requires thyroid function test review by study physician (SP) to determine eligibility)
17. Recent weight loss (more than or equal to 5% body weight) in the past 3 months

    * Participants presenting with systolic blood pressure (SBP) greater than 159 mmHg and/or diastolic blood pressure (DBP) greater than 99 mmHg at the Intake visit will be instructed to sit quietly for 10 minutes. Then the participant will have a second blood pressure reading taken after a 10 minute period. If, after the second reading the SBP greater than 159 mmHg and the DBP greater than 99 mmHg, the individual will be instructed to sit comfortably for 10 minutes and then have a third blood pressure reading. If, after the third reading the SBP greater than 159 mmHg and the DBP greater than 99 mmHg, the individual will be ineligible to participate.

Medications:

1. Current or recent use (last 14 days) of weight loss medication, and/or use of medications known to impact weight (e.g. corticosteroids, excluding inhaled).

General Exclusion:

1. Current, anticipated, or pending enrollment in another research program over the next 2-3 months that could potentially affect subject safety and/or the study data/design as determined by the Principal Investigator and/or Study Physician.
2. Not planning to live in the area for the next 9 months.
3. Previous participation in this trial (i.e., previously randomized and started study medication).
4. Any impairment (physical and/or neurological) including visual or other impairment preventing ability to complete study tasks.
5. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca L Ashare, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Smoking Cessation Counseling & Liraglutide | Smoking Cessation Counseling & Placebo
Started | 19 | 21
Completed | 5 | 9
Not Completed | 14 | 12
Not completed — Lost to Follow-up | 3 | 7
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smoking Cessation Counseling & Liraglutide | Smoking Cessation Counseling & Placebo | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 21 | 38
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (6.2) | 56.4 (5.6) | 57.2 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 18 | 21 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 12 | 21
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 21 | 40
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 36.9 (1.8) | 35.8 (1.4) | 36.3 (1.1)
Cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes] | 16.6 (2.1) | 16.7 (1.8) | 16.7 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 7-day Point Prevalence Smoking Abstinence at 12 Weeks Post-Target Quit Date
Description: Biochemically verified carbon monoxide (CO) reading <5 using a Vitalograph Breath CO Analyzer
Time Frame: Week 18
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Counseling & Liraglutide | Smoking Cessation Counseling & Placebo
Number analyzed (Participants) | 19 | 21
Participants | 2 | 2

2. Primary Outcome: Number of Participants With 7-day Point Prevalence Smoking Abstinence at 26 Weeks Post-Target Quit Date
Description: Biochemically verified carbon monoxide (CO) reading <5 using a Vitalograph Breath CO Analyzer
Time Frame: Week 32
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Counseling & Liraglutide | Smoking Cessation Counseling & Placebo
Number analyzed (Participants) | 19 | 21
Participants | 2 | 2

3. Secondary Outcome: Body Weight at 12 Weeks Post-Target Quit Date
Description: Body weight will be measured by digital scale (pounds, ounces) wearing light clothing without shoes
Time Frame: Week 18
Population: The number analyzed reflects rates due to attrition as only those who completed visits could provide measurement.
Measure: Mean (Standard Deviation); unit: lb
Arm/Group | Smoking Cessation Counseling & Liraglutide | Smoking Cessation Counseling & Placebo
Number analyzed (Participants) | 3 | 8
lb | 209.8 (14.4) | 212.6 (17.8)

4. Secondary Outcome: Body Weight at 26 Weeks Post-Target Quit Date
Description: Body weight will be measured by digital scale (pounds, ounces) wearing light clothing without shoes
Time Frame: Week 32
Population: The number analyzed reflects rates due to attrition as only those who completed visits could provide measurement.
Measure: Mean (Standard Deviation); unit: lb
Arm/Group | Smoking Cessation Counseling & Liraglutide | Smoking Cessation Counseling & Placebo
Number analyzed (Participants) | 2 | 7
lb | 234.4 (37.6) | 209.8 (19.0)

5. Other Pre Specified Outcome: Calories Consumed Per Day
Description: The research team staff will use a multi-pass method with an interactive computerized software program, the Automated Self-Administered 24-hour Recall (ASA24®) tool to determine total kcal/day with participants over the phone.
Time Frame: Weeks 0, 5, 18, & 32
Population: The number analyzed differs due to attrition. Only those who completed each visit were analyzed.
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Smoking Cessation Counseling & Liraglutide | Smoking Cessation Counseling & Placebo
Number analyzed (Participants) | 19 | 21
kcal/day
  Week 0 | 1994.4 (680.7) | 1703.9 (484.7)
  Week 5: number analyzed (Participants) | 15 | 17
  Week 5 | 1572.2 (563.7) | 1781.3 (662.9)
  Week 18: number analyzed (Participants) | 5 | 10
  Week 18 | 1352.1 (485.2) | 1582.6 (494)
  Week 32: number analyzed (Participants) | 5 | 8
  Week 32 | 1360.3 (405.0) | 1797.6 (518.5)

ADVERSE EVENTS:
Time Frame: 8 months
Description: The definitions do not differ. Adverse event reporting was completed using a symptom checklist, listing all expected side effects for the study drug, which was administered at all study visits and included severity rating and description of the symptom. Participants were also given the opportunity to report any events that were not listed on the checklist, provide a severity rating and description.
Arm/Group | Smoking Cessation Counseling & Liraglutide | Smoking Cessation Counseling & Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 2/21
Other Adverse Events (participants affected / at risk) | 18/19 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smoking Cessation Counseling & Liraglutide (N=19) | Smoking Cessation Counseling & Placebo (N=21)
Pain (General disorders) | 0 (0) | 1 (1)
TIA (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Smoking Cessation Counseling & Liraglutide (N=19) | Smoking Cessation Counseling & Placebo (N=21)
Acid Reflux (Gastrointestinal disorders) | 5 | 4
Abdominal Pain (Gastrointestinal disorders) | 4 | 4
Anxiety (Psychiatric disorders) | 4 | 8
Belching (Gastrointestinal disorders) | 4 | 2
Bloating (Gastrointestinal disorders) | 1 | 4
Bruising at injection site (Skin and subcutaneous tissue disorders) | 4 | 4
Constipation (Gastrointestinal disorders) | 10 | 4
Decreased Appetite (Gastrointestinal disorders) | 15 | 13
Diarrhea (Gastrointestinal disorders) | 6 | 3
Dizziness (General disorders) | 6 | 6
Dry Mouth (General disorders) | 5 | 10
Fatigue (General disorders) | 11 | 9
Flatulence (Gastrointestinal disorders) | 5 | 5
Headache (General disorders) | 9 | 12
Hypertension (Cardiac disorders) | 7 | 12
Indigestion (Gastrointestinal disorders) | 5 | 2
Insomnia (General disorders) | 7 | 10
Nausea (Gastrointestinal disorders) | 12 | 8
Vomiting (Gastrointestinal disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT03712098/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT03712098/ICF_002.pdf